CLINICAL TRIAL: NCT03187704
Title: Boston Puerto Rican Health Study - Project 4
Brief Title: Boston Puerto Rican Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Doug Brugge, Professor, Tufts University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: BPRHS-Project4
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Air Pollution; Cardiovascular Health
Keywords: air filtration, HEPA, In-home,

STUDY DESIGN:
Intervention Model Description: Randomized cross-over
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were blinded as to filtration and no filtration. The lab was blinded as to which samples were from filtration or no filtration periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- filtration (Active Comparator): Air filtration in homes
  Interventions: Other: HEPA air filtration
- no filtration (Sham Comparator): Sham air filtration
  Interventions: Other: HEPA air filtration

INTERVENTIONS:
Other: HEPA air filtration — Air filters were placed in participant homes

SUMMARY:
The study is a blinded cross over test of in-home air filtration. Participants will have a window unit air filter (HEPA) installed that will filter for 3 weeks and do sham filtration for another 3 weeks. During the time that the filter is installed in the home a machine that measures particulate air pollution of the type that the filter is designed to remove will be installed. A survey will be administered, blood samples taken and blood pressure measured immediately prior to starting the filter, at 3 weeks when the filtration is changed from sham to real filtration or visa versa and at the end of the second three week period. All participants will be recruited from the Boston Puerto Rican Health Study cohort.

DETAILED DESCRIPTION:
Project 4 Protocol:

I. Aims and Hypotheses

H1: That in-home active HEPA filtration will reduce ultrafine particle (UFP) levels >70% compared to sham filtration. Further, that HEPA filtration will reduce all size classes of ultrafine particles equally well.

H2: That markers of cardiovascular health, including C-reactive protein, fibrinogen, IL-6 and tumor necrosis factor alpha receptor, will be lower after living with active HEPA filtration compared to sham filtration.

H3: In-home HEPA filtration will be seen by policy-makers as an effective policy option for reducing UFP exposure in near-highway residences.

The study was a double-blind, randomized crossover trial in which each participant served as their own control, thereby greatly reducing the role of time-invariable confounders. Up to two homes were enrolled and randomized at a time, with one allocated to receive HEPA filtration and the other sham filtration first. At three weeks, the homes were switched from HEPA filtration to sham or vice versa. There was no washout period between sham and HEPA filtration. While field staff were aware of the type of filter in use, the participants and the lab that analyzed blood samples were not. The approach and methods were largely similar to another HEPA intervention we conducted in public housing in the City of Somerville, which was still in progress at the start of this study.

Participants were recruited from the BPRHS cohort. The parent study was in the process of follow-up at approximately five years since baseline with close to 1000 participants remaining. The cohort staff recommended non-smoking participants who they thought might be receptive to our intervention. Of the 25 participants enrolled, 23 (92%) completed the study and were included in the analysis. One home was removed due to the failure of the flow sensor, which identified indoor versus outdoor air, while the other was removed because the participant opted to end the study early. All participants lived in the cities of Boston or Chelsea. Data on demographics and health were obtained from surveys collected during longitudinal follow-up of the cohort. For the participants receiving the intervention, the investigators collected additional surveys with information on recent exposures, recent illnesses, and participant time-activity patterns (at home, work/school, travel on highways, other).

Participants signed consent forms for the parent study and a separate consent for the air filtration intervention. The studies were approved by the IRBs at Tufts Medical Center, Northeastern University, and the University of Massachusetts Lowell.

The intervention Window-mounted HEPAirX air filtration units (Air Innovations, Inc., North Syracuse, NY, USA) equipped with MERV 17 filters (rated to remove ≥99.97% of particles ≥0.3 μm in diameter) were used. These units can operate at ~10 exchanges/hour in a 28.3 m3 (103 ft3) room and have user-controlled air heating and cooling elements. The units were installed preferentially in living rooms of apartments (N=16), where participants spent much of their day. Eight units were installed in bedrooms due to space restrictions or because living room windows did not accommodate the HEPAirX unit. To maximize particle removal, the HEPA units were operated at the highest possible fan speed and the vents were blocked so that there was no flow of outdoor air through the unit into the apartment. Also, participants were asked to keep windows closed as much as possible during the study period to minimize infiltration from outside. Filters were changed in each apartment after 21 days (HEPA for sham or vice versa). A new HEPA filter (MERV 17) was used in each apartment. The sham filter was an empty, perforated sheet metal box that was the same size and shape and had the same appearance as the metal frame around the HEPA filters. The HEPAirX sounded the same regardless of sham or HEPA filtration. A sign written in English and Spanish was placed on the HEPA-unit cover asking participants not to tamper with or expose the filter.

Air pollution monitoring Particle number concentrations (PNC) were measured continuously during the six-week trial in each apartment using water-based condensation particle counters (CPC; TSI Model 3783, d50 7 nm, maximum detectable particle >3 µm). The CPCs were installed in the same room as the HEPAirX unit and recorded 30-second mean PNC (one-minute mean PNC in the first five homes). Both outdoor and indoor PNC were measured; a solenoid valve switched every 15 minutes between two, 1-m-long conductive silicon inlet tubes: one pulled from indoors and the other pulled from outdoors. An in-line flow sensor logged different voltages depending on whether a flow was detected in the line (2.49 V with flow, ~1.00 V with no flow); these were used to identify indoor and outdoor sampling periods. Before the start of the intervention in each apartment, CPC flow rates were measured using a flow meter (TSI Model 4140) (no discrepancies were observed throughout the study). The CPC vacuum was also checked for leaks by placing a polyethersulfone membrane filter (rated at 99.96% removal efficiency for 0.45 µm particles) on the inlet to insure the CPC measured <100 particles/cm3. Sites were visited weekly for regular maintenance (flow checks, time resets, etc.) and to download data. Data flagged by the CPC as erroneous (typically <1% of all data per home) were removed from the data set. Consistent with manufacturer specifications, all CPCs performed within 10% of one another in laboratory side-by-side comparisons.

The Somerville study, which the investigators combined with the current study in a meta-analysis, followed the same study design and methods with the following differences: 1) there was no outdoor monitoring; 2) all study participants resided within 200 m of a highway; and 3) the study participants differed in their demographics.

Indoor sources Indoor measurements reflect both the fraction of outdoor UFP that infiltrate indoors and indoor-generated UFP - e.g., from cooking, candle and incense burning, and cleaning. These sources result in large but variable magnitude spikes in indoor concentrations and further, the rate of decay of these spikes depends on several factors, such as source strength and duration, room volume and ventilation rate. It is thus challenging to completely separate the contributions from outdoor and indoor UFP sources based on indoor PNC measurements. Nonetheless, to test effects of indoor spikes on associations with biomarkers, the investigators generated a PNC time-series for each home and calculated the six-hour moving median for indoor PNC measurements. The investigators then calculated the standard deviation for the three-week period corresponding to HEPA or sham filtration; indoor measurements that were two standard deviations above this six-hour moving median were classified as spikes and replaced with the last indoor measurement that was not considered to be a spiked value. Even though the investigators' method did not completely remove the contribution from indoor sources, it attenuated the contributions from spikes that skewed the three-week indoor average values used as exposure concentrations.

Biomarkers A venous blood sample was collected at the start, at the change of filter types (end of week 3) and at end of the intervention (end of week 6). Samples were transported to the Human Nutrition Research Center on Aging (Tufts University, Boston campus), where they were processed to plasma and stored at minus 80 ºC within 1-3 h of collection. Participants were instructed to fast overnight prior to the blood draws (79% confirming fasting), which occurred between 8 and 10 AM. Samples were assayed in batches using immunoassay kits for TNF-RII (Quantitative, R&D Systems, Minneapolis, MN, USA) and IL-6 (Quantitative HS, R&D Systems). High sensitivity CRP (hsCRP) was measured by a solid-phase, two-site chemiluminescent immunometric assay, (IMMULITE 2000, Siemens Healthcare Diagnostics, Los Angeles, CA 90045). These biomarkers are a measure of the levels of systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the larger parent cohort of the BPRHS

Exclusion Criteria:

* None since already enrolled in the cohort

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Blood biomarkers | 6 weeks
  hsCRP, IL-6, TNFRII

CONTACTS AND LOCATIONS:
Overall Officials: Doug Brugge, PhD, Study Director — Tufts University
Locations (1):
- Tufts University School of Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data

REFERENCES:
- [Background] Padro-Martinez LT, Owusu E, Reisner E, Zamore W, Simon MC, Mwamburi M, Brown CA, Chung M, Brugge D, Durant JL. A Randomized Cross-over Air Filtration Intervention Trial for Reducing Cardiovascular Health Risks in Residents of Public Housing near a Highway. Int J Environ Res Public Health. 2015 Jul 10;12(7):7814-38. doi: 10.3390/ijerph120707814. PMID 26184257
- [Background] Bhangar S, Mullen NA, Hering SV, Kreisberg NM, Nazaroff WW. Ultrafine particle concentrations and exposures in seven residences in northern California. Indoor Air. 2011 Apr;21(2):132-44. doi: 10.1111/j.1600-0668.2010.00689.x. Epub 2010 Oct 28. PMID 21029183
- [Background] Rim D, Wallace L, Persily A. Infiltration of outdoor ultrafine particles into a test house. Environ Sci Technol. 2010 Aug 1;44(15):5908-13. doi: 10.1021/es101202a. PMID 20666560
- [Background] Wallace L, Kindzierski W, Kearney J, MacNeill M, Heroux ME, Wheeler AJ. Fine and ultrafine particle decay rates in multiple homes. Environ Sci Technol. 2013 Nov 19;47(22):12929-37. doi: 10.1021/es402580t. Epub 2013 Nov 6. PMID 24143863
- [Background] Beko G, Weschler CJ, Wierzbicka A, Karottki DG, Toftum J, Loft S, Clausen G. Ultrafine particles: exposure and source apportionment in 56 Danish homes. Environ Sci Technol. 2013 Sep 17;47(18):10240-8. doi: 10.1021/es402429h. Epub 2013 Sep 4. PMID 23957328